CLINICAL TRIAL: NCT06916910
Title: Analysis of Predictive Factors for Urinary Leakage After Partial Nephrectomy for Renal Hilum Tumors: A Multicenter Retrospective Clinical Study
Brief Title: Analysis of Predictive Factors for Urinary Leakage After Partial Nephrectomy for Renal Hilum Tumors
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Collaborators: The Second Affiliated Hospital of Fujian Medical University (Other); The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: MRCTA,ECFAH OfFMU[2024]905
Record Dates: First submitted 2025-02-24; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Partial Nephrectomy; Renal Hilum Tumors; Urinary Leakage
Keywords: urinary leakage; partial nephrectomy; renal hilum tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we plan to explore the risk factors closely related to the occurrence of urinary leakage after partial nephrectomy for renal hilum tumors through retrospective analysis of multicenter clinical data, thereby providing clinical guidance value for the prevention of postoperative urinary leakage.

ELIGIBILITY:
Inclusion Criteria:

* CT or MRI angiography indicates a renal hilum tumor, and the patient has undergone partial nephrectomy;
* The Eastern Cooperative Oncology Group (ECOG) performance status score is between 0 and 1, and the age is between 18 and 75 years old;
* The clinicopathological data are complete;
* There is no infection, autoimmune disease, hematological disease, or other malignancies.

Exclusion Criteria:

* The patient has surgical contraindications;
* There are congenital malformations of the urinary system, obstructive nephropathy, or other diseases that seriously affect the function of the urinary system before surgery;
* The patient has received relevant treatments that may affect the results of this study, such as radiotherapy in the kidney area, a history of kidney surgery, etc.;
* There are tumors in both kidneys.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing partial nephrectomy for renal hilum tumors
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-09-18 (Estimated); Study Completion 2025-09-18 (Estimated)

PRIMARY OUTCOMES:
Postoperative urinary leakage | the postoperative perirenal drainage volume being greater than 50 ml for 7 consecutive days and the creatinine level of the drainage fluid being similar to that of urine(μmol/L), or postoperative urinary leakage being suspected by imaging examination.
  Postoperative urinary leakage is defined as the postoperative perirenal drainage volume being greater than 50 ml for 7 consecutive days and the creatinine level of the drainage fluid being similar to that of urine(μmol/L), or postoperative urinary leakage being suspected by imaging examination.

CONTACTS AND LOCATIONS:
Locations (1):
- first hospital affiliated of Fujian medical university, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided